CLINICAL TRIAL: NCT03147586
Title: Influence of Immune Nutrition Diet on 90-Day Outcomes in Patients Undergoing Radical Cystectomy and Bladder Substitutions: A Randomized Controlled Trial
Brief Title: Influence of Immune Nutrition Diet on 90-Day Outcomes in Patients Undergoing Radical Cystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hossam Nabeeh, Msc, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD/16.10.55
Record Dates: First submitted 2017-03-12; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Bladder Cancer; Oncology; Infection; Complication; Muscle Invasive; Radical Cystectomy
Keywords: Immune Nutrition; Morbidity
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms; Infections | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bio-tech and omega-3 plus (Active Comparator): Bio-tech (Biopharm pharmaceutical) powder 30 mg t.d.s. (contains multivitamins and essential amino acids) plus omega-3 plus (SEDICO pharmaceutical) capsules t.d.s (source for omega-3 fatty acids) 1 week before and 2 week after surgery
  Interventions: Drug: Bio-tech and omega-3 plus
- placebo (Placebo Comparator): placebo powder 30 mg t.d.s plus placebo capsules t.d.s for 1 week before and 2 week after surgery
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bio-tech and omega-3 plus — immune nutrition : Bio-tech ( multivitamins and essential amino acids), and omega-3 plus (omega-3 fatty acids)
  Arms: Bio-tech and omega-3 plus
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This is a randomised double-blinded placebo-controlled phase IV trial with two parallel treatment groups receiving either immune nutrition diet (IND) or conventional diet for 2weeks peri-radical cystectomy. Patients will be stratified according to the gender, body mass index, and the type of urinary diversion (orthotopic neobladder or ileal conduit). The primary end-point is to determine, in intention to treat analysis, the influence of IND on 90-day postoperative morbidity. Secondary study end-points will be the effect of IND on infectious as well as non-infectious complications over 90 days, compliance and adverse effects of IND. Finally, an ancillary study will be performed to evaluate whether the IND costs could counterbalance, by its benefits, the health care costs.It is envisaged to finish patients' recruitment within 24 months

DETAILED DESCRIPTION:
Radical cystectomy (RC) with pelvic lymphadenectomy is established as the gold standard surgical treatment of muscle invasive bladder cancer. Major complication rates at 90 days as high as 25% have been reported using a standardized reporting methodology even with the use of enhanced recovery protocol after surgery (ERAS), high lighting the significance of identification of the potential predictors to alleviate patients suffering after this complex procedure.

A major preoperative potentially reversible risk factor for severe postoperative morbidity is nutritional status, even; it is considered recently the missed ring in the all available morbidity prognostic indices. This was typically proving in other kinds of cancer. For instance, it has been shown that patients at nutritional risk have had significantly postoperative complications 10% as high as compared to those not at nutritional risk as well as elevated rates of anastomotic leak and infections after colorectal surgery. Likewise, in an observational trial, there was an increased risk of postoperative complications in malnourished patients undergoing pneumonectomy for lung cancer.Furthermore, the hazardous impact of malnutrition does extend beyond the potential morbidity to increased cost, hospital stay, and readmission rates. Not surprisingly, the prognostic nutritional index was shown, additionally, to influence the survival after total gastrectomy for patients with gastric cancer.

With respect to urological literature, the incidence of malnutrition amany surgical candidates largely differs according to the methodology implicated, ranging from 26-43% according to the nutritional index scoring system and 19% using serum albumin level and weight loss and body mass index. Moreover, the influence of poor nutritional status on postoperative morbidity has been clearly identified.

Johnson et al have demonstrated an increased incidence of postoperative complications from 55% to 67% for patients with nutritional deficiency portrayed by low serum albumin level. Similarly yet in gynecological cancers, hypoalbuminemia was an independent surrogate for adverse postoperative events. Therefore, it has been highly recommended to implicate innovative nutritional interventions for optimizing the outcome after radical cystectomy.What is worth mention is that the active ingredients of immune diet were considerably the same across studies on different cancers, and principally including arginine, omega-3 fatty acids, and glutamine which have been proved to ameliorate the inflammatory and stress response of the body to surgery, and consequently, minimizing the postoperative morbidity. It is also particularly important to note that oral diet had been valued over parenteral injections concerning efficacy and safety.

To date, only two pilot trials have been applied elucidating the beneficial effect of immune nutrition diet (IND) on postoperative morbidity and surgery-induced inflammations after radical cystectomy.Hamilton-Reeves and associates have represented a reduction of 33% and 39% in overall complications and infection rates, respectively. Then again, the authors have shown a potential effect of the IND on the laboratory markers of inflammation. Equally important, a decline by just below the half, falling from 77% to 40% complications rate, and by more than half, from 66% to 20% infection rate, were noted in a prospective cohort compared with historical control.

Yet, these studies were limited by the relative-low number of patients as both were considered "pilot". In addition, neither of both studies had determined the nutritional status of the candidates prior to enrolment in the study protocol. Furthermore, there was no control for some confounding variables like gender, body mass index and type of diversion, which definitely would affect the primary outcome of these studies.

In this context, this protocol was designed to assess the impact of IND on patients undergoing radical cystectomy controlling for every single potential confounding variable.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bladder cancer eligible for radical cystectomy and urinary diversions
* Willing to be randomized

Exclusion Criteria:

* Non-compliance and /or allergy with oral nutrition diet.
* Non-organ confined disease
* Associated comorbidities e.g. Gout and Rheumatoid arthritis
* Weight loss more than10% (with respect to usual body weight) in the past 6 months
* Hepatic dysfunction (Child-Pugh class more than B), and renal dysfunction (serum creatinine level more than3 mg/dL, hemodialysis),
* Untreated infections
* Immune disorders.
* Chronic gastrointestinal tract disease eg.crohn's disease or previous surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-10-30 (Estimated); Study Completion 2017-10-30 (Estimated)

PRIMARY OUTCOMES:
The overall 90-day postoperative complication between groups measured by modified Dindo-Clavien system | 3 months
  measured by modified Dindo-Clavien system

SECONDARY OUTCOMES:
The effect of immune nutrition diet on nutritional status of radical cystectomy patients measured by validated nutritional assessment scores | 3 months
  measured by validated nutritional assessment scores
The effect of immune nutrition diet on anthropometric measures of radical cystectomy patients measured by skinfold thickness in centimetres | 3 months
  measured by skinfold thickness in centimetres

CONTACTS AND LOCATIONS:
Overall Officials: Atallah A. Shaaban, MD, Study Chair — Urology and nephrology center; Hassan Abo-Elenin, MD, Study Director — Urology and nephrology center; Ahmed Mosbah, MD, Study Director — Urology and nephrology center; Ahmed Harraz, MD, Principal Investigator — Urology and nephrology center; Abdelwahab R. Hashem, Msc, Principal Investigator — Urology and nephrology center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
meta-analyses by contact the Prof. Atallah Ahmed Shaaban MD (Study Chair)